CLINICAL TRIAL: NCT05152160
Title: Clinical Trial of Umbilical Cord Mesenchymal Stem Cells in the Treatment of Moderate/Severe Chronic Graft-versus-host Disease
Brief Title: Umbilical Cord Mesenchymal Stem Cells in the Treatment of Moderate/Severe Chronic Graft-versus-host Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen University General Hospital (Other)
Responsible Party: Principal Investigator, YuLi, Professor, Shenzhen University General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEM-ONCO-014
Record Dates: First submitted 2021-11-22; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-08

CONDITIONS: Graft Vs Host Disease
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Umbilical Cord Mesenchymal Stem Cell Therapy
  Interventions: Biological: Umbilical Cord Mesenchymal Stem Cell Therapy

INTERVENTIONS:
Biological: Umbilical Cord Mesenchymal Stem Cell Therapy — Umbilical Cord Mesenchymal Stem Cell Therapy

SUMMARY:
cGVHD is a systemic disease with multi-system damage similar to autoimmune and other immune diseases. It can affect multiple organs such as skin, liver, kidney, and peripheral nerves, causing a serious decline in the quality of life of patients, and death in the late stage of transplantation. According to the cGVHD prognostic risk scoring system (revised Risk Group) revised by the European Society for Blood and Bone Marrow Transplantation (EBMT) in 2017, the 3-year survival rate of patients with rRG1 (0-3 points) is about 93.3 ± 6.4%, and rRG2 (4-6 points) about 84.9 ± 3.4%, rRG3 (7-9 points) about 70.9 ± 4.4%, rRG4 (≥10 points) about 32.0 ± 1.1%, it can be seen that moderate to severe cGVHD directly affects the survival of allo-HSCT patients.

Once moderate or severe cGVHD is diagnosed, glucocorticoids with or without calcineurin inhibitor (CNI) are first-line drugs, but the effective rate is less than 50%, and the prognosis of hormone-resistant severe cGVHD is extremely poor even if second-line treatment is added. Second-line treatments include monoclonal antibodies, immunosuppressants, chemotherapy drugs, phototherapy or others. Most of them cannot improve the long-term survival rate. The main reason is that these treatments suppress immunity for a long time, which increases the risk of infection and reduces the survival rate. In this context, the treatment of mesenchymal stromal stem cells (MSCs) provides a new path for clinical treatment of cGVHD.

DETAILED DESCRIPTION:
Chronic graft-versus-host disease (cGVHD) refers to the clinicopathological synthesis of lymphocytes from the donor attacking the recipient's organs during the process of rebuilding the donor's immunity after allogeneic hematopoietic stem cell transplantation (allo-HSCT) Signs (including classic cGVHD and overlap syndrome) are one of the main complications after transplantation, with an incidence of 30% to 70%. cGVHD is a systemic disease with multi-system damage similar to autoimmune and other immune diseases. It can affect multiple organs such as skin, liver, kidney, and peripheral nerves, causing a serious decline in the quality of life of patients, and death in the late stage of transplantation. main reason. According to the cGVHD prognostic risk scoring system (revised Risk Group) revised by the European Society for Blood and Bone Marrow Transplantation (EBMT) in 2017, the 3-year survival rate of patients with rRG1 (0-3 points) is about 93.3 ± 6.4%, and rRG2 (4-6 points) About 84.9 ± 3.4%, rRG3 (7-9 points) about 70.9 ± 4.4%, rRG4 (≥10 points) about 32.0 ± 1.1%, it can be seen that moderate to severe cGVHD directly affects the survival of allo-HSCT patients.

Once moderate or severe cGVHD is diagnosed, glucocorticoids with or without calcineurin inhibitor (CNI) are first-line drugs, but the effective rate is less than 50%, and the prognosis of hormone-resistant severe cGVHD is extremely poor even if second-line treatment is added. Second-line treatments include monoclonal antibodies, immunosuppressants, chemotherapy drugs, phototherapy or others. Most of them cannot improve the long-term survival rate. The main reason is that these treatments suppress immunity for a long time, which increases the risk of infection and reduces the survival rate. In this context, the treatment of mesenchymal stromal stem cells (MSCs) provides a new path for clinical treatment of cGVHD.

In 2002, Frassoni reported for the first time that MSCs expanded in vitro were used to evaluate the efficacy of allo-HSCT. Allo-HSCT transplanted patients with hematological malignancies were enrolled. MSCs were derived from the donor's bone marrow. After expanded in vitro, participants were combined with the donor's hematopoietic stem cells for reinfusion. As a result, the incidence of aGVHD in the MSCs expansion group and cGVHD within 6 months was significantly lower in the control group, the 6-month OS was significantly higher than that in the control group, and there was no significant difference in the recurrence rate. Subsequently, in 2004, Le Blanc and others successfully used third-party MSCs to successfully treat a refractory grade IV intestinal combined with liver aGVHD for the first time. Subsequently, MSCs were increasingly used in clinical studies for the treatment of GVHD. More clinical trials have shown that umbilical cord-derived MSCs cultured in vitro can not only promote the implantation of hematopoietic stem cells (HSC), but also reduce the incidence of severe GVHD in patients, showing a good therapeutic effect.

ELIGIBILITY:
Inclusion Criteria:

1. Age 14-70 (≥14, ≤70) one year old, no gender limit;
2. The subject voluntarily participates in the study, and he or his legal guardian signs the "Informed Consent";
3. CGVHD occurred after transplantation of allogeneic hematopoietic stem cells (umbilical cord blood, bone marrow or mobilized peripheral blood) with the primary disease of hematological malignancy, and was diagnosed as moderate/severe cGVHD according to the "Chinese Expert Consensus on the Diagnosis and Treatment of cGVHD (2021 Edition)";
4. Those who are tolerant to the first-line standard treatment regimen (glucocorticoid with or without calcineurin inhibitor):

1) The organ damage that has been involved in the past is aggravated; 2) People with new organ involvement; 3) No improvement in symptoms and signs after 1 month of regular medication (such as glucocorticoid therapy alone, progress in the initial 2 weeks, no improvement in 6-8 weeks, consider glucocorticoid resistance); 4) At 2 months, prednisone cannot be reduced to less than 1.0mg/kg/d; 5. EOCG score ≤ 3 points.

Exclusion Criteria:

-

Patients with any of the following cannot be included in this study:

1. Serum virological examination showed that hepatitis C virus (HCV) antibody, Treponema pallidum (TP) antibody or human immunodeficiency virus (HIV) antibody test results were positive;
2. People with severe hepatic vein occlusive disease or sinus vein occlusive syndrome;
3. According to the evaluation of the investigator, patients with cytomegalovirus (CMV) enteritis, transplantation-related thrombotic microangiopathy (TA-TMA), and gastrointestinal infections caused by diarrhea cannot be ruled out clinically; the pathological diagnosis criteria of CMV enteritis are: intestinal mucosa. Large cells of basic inclusion bodies, immunohistochemical CMV early/late antigen positive, intestinal mucosal homogenate CMV nucleic acid PCR positive;
4. Patient renal function: creatinine clearance rate <30mL/min; creatinine clearance rate is calculated by Cockcroft-Gault formula: Ccr(ml/min)=[(140-age)×weight (kg)]/(72×serum creatinine( mg/dL), for women, according to the calculation result × 0.85), the unit of creatinine should be paid attention to during the calculation of creatinine clearance;
5. Within 6 months before enrollment, there is evidence that the patient has other diseases or their physiological conditions may interfere with the evaluation results of this test, or the complications are severely life-threatening, including but not limited to uncontrolled infections, pulmonary hypertension, severe Cardiac insufficiency (NYHA class III and IV), unstable angina or acute myocardial infarction, refractory hypertension (defined as the simultaneous use of 3 different types of antihypertensive drugs [one of which is a diuretic] Higher than 180/110mmHg) (subject to the diagnosis of hospitalized medical records), etc.;
6. Patients with active malignant solid tumors within the first 5 years of the study, except for radically cured cervical cancer, in situ localized prostate cancer and non-melanoma skin cancer;
7. Patients with myelofibrosis;
8. People who suffer from mental or neurological diseases and cannot express their wishes correctly;
9. Those who have a history of severe allergies to blood components or blood products, or those who have a history of allergies to heterologous proteins;
10. Breastfeeding women, or female patients who have pregnancy plans or egg donation plans from the start of the study to the follow-up period, and male patients (or their partners) have birth plans or sperm donation plans from the start of the study to the follow-up period, and are unwilling to take contraceptive measures ；
11. Those determined by the investigator to be unsuitable to participate in this clinical trial;
12. Those who have participated in other clinical trials within the previous month.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Disease-related clinical reactions | Change frome baseline clinical manifestationc of cGVHD at 8 weeks
  Complete remission, partial remission, disease progression

SECONDARY OUTCOMES:
PFS | From admission to the end of follow up, up to 2 years.
  Progression-Free-Survival

CONTACTS AND LOCATIONS:
Overall Officials: Li Yu, Dr, Principal Investigator — Shenzhen University General Hospital
Locations (1):
- Li Yu, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No